CLINICAL TRIAL: NCT03577574
Title: A Prospective, Randomised, Single-masked Comparison of Retrobulbar Anesthesia, Peribulbar Anesthesia and Topical Combined Subconjunctival(Two-step) Anesthesia in Posterior Vitrectomy
Brief Title: Study of Two-step Anesthesia in Posterior Vitrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SHIRB2018013
Record Dates: First submitted 2018-05-28; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- retrobulbar anesthesia group (Active Comparator): 2% lidocaine 4ml injected into retrobulbar space
  Interventions: Procedure: retrobulbar anesthesia
- peribulbar anesthesia group (Active Comparator): 2% lidocaine 4 to 8ml injected into peribulbar space
  Interventions: Procedure: peribulbar anesthesia
- two step anesthesia group (Experimental): conjunctival cul-de-sac anesthetized with 0.5% proparacaine hydrochloride drops three times + 2% lidocaine 0.6 to 0.8ml subconjunctival injection
  Interventions: Procedure: two step anesthesia

INTERVENTIONS:
Procedure: retrobulbar anesthesia — 2% lidocaine 4ml injected into retrobulbar space
  Arms: retrobulbar anesthesia group
Procedure: peribulbar anesthesia — 2% lidocaine 4 to 8ml injected into peribulbar space
  Arms: peribulbar anesthesia group
Procedure: two step anesthesia — conjunctival cul-de-sac anesthetized with 0.5% proparacaine hydrochloride drops three times + 2% lidocaine 0.6 to 0.8ml subconjunctival injection
  Arms: two step anesthesia group

SUMMARY:
A prospective, randomised, single-masked comparison of local anaesthetic approaches including topical anesthesia combined sub-conjunctival anesthesia(two-step anesthesia) for minimally invasive vitrectomy（TAMIV）vs peribulbar block vs retrobulbar block

DETAILED DESCRIPTION:
Purpose: topical anesthesia combined sub-conjunctival anesthesia(two-step anesthesia) for minimally invasive vitrectomy Methods: This prospective, randomized, single-blinded clinical trail is conducted at Shanghai Aier Eye Hospital. Selected group of 60 patients with retinal-vitreous diseases will be randomized divided into 3 groups and underwent 25-gauge vitrectomy. Group1 uses two-step anesthesia , whereas Group 2 uses retrobulbar anesthesia, group 3 uses peribulbar anesthesia. A 5-point Visual Analogue Pain Scale is used to assess patients' pain score and surgeon's ease while operating. Any complications therefore will be made note of.

ELIGIBILITY:
Inclusion Criteria:

* Proliferative diabetic retinopathy (PDR);
* Vitreous haemorrhage (VH);
* Retinal detachment (RD);
* Retinal vein occlusion(RVO);
* Other diseases (idiopathic macular hole, macular pucker and high myopic maculopathy);
* Silicone oil-filled eye.

Exclusion Criteria:

* Communication problems;
* Allergy to amide-type local anaesthetic agents;
* History of vitreoretinal surgery or orbital surgery;
* Orbital deformity;
* With episcleral adjunct surgery;
* Trauma;
* Keratitis;
* Conjunctivitis and active uveitis.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-02 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
pain scores | During surgery
  5-point Visual Analogue Pain Scale(VAPS): Grade 1: No pain or discomfort; Grade 2: mild pain or discomfort; Grade 3: moderate pain or discomfort; Grade 4: severe pain or discomfort;

SECONDARY OUTCOMES:
surgeon's ease | During surgery
  Grade 1: No discomfort; Grade 2: mild discomfort; Grade 3: moderate discomfort; Grade 4: severe discomfort;

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Study Director — Shanghai Aier Eye Hosptial
Locations (1):
- Wensheng Li, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan WM, Loo AV, Tam BS. Topical anesthesia in posterior vitrectomy. Retina. 2000;20(5):563-5. doi: 10.1097/00006982-200005000-00029. No abstract available. PMID 11039443
- [Background] Bahcecioglu H, Unal M, Artunay O, Rasier R, Sarici A. Posterior vitrectomy under topical anesthesia. Can J Ophthalmol. 2007 Apr;42(2):272-7. PMID 17392852
- [Background] Schrader WF, Schargus M, Schneider E, Josifova T. Risks and sequelae of scleral perforation during peribulbar or retrobulbar anesthesia. J Cataract Refract Surg. 2010 Jun;36(6):885-9. doi: 10.1016/j.jcrs.2009.12.029. PMID 20494757
- [Background] Takaschima A, Marchioro P, Sakae TM, Porporatti AL, Mezzomo LA, De Luca Canto G. Risk of Hemorrhage during Needle-Based Ophthalmic Regional Anesthesia in Patients Taking Antithrombotics: A Systematic Review. PLoS One. 2016 Jan 22;11(1):e0147227. doi: 10.1371/journal.pone.0147227. eCollection 2016. PMID 26800356